CLINICAL TRIAL: NCT00094055
Title: Phase 2 Study of the Anti-Angiogenesis Agent AG-013736 in Patients With Metastatic Thyroid Cancer Who Are Refractory to or Not Suitable Candidates for 131 I Treatment
Brief Title: Study of the Anti-angiogenesis Agent AG-013736 in Patients With Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061014
Record Dates: First submitted 2004-10-08; First posted 2004-10-11 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axitinib [AG-013736] (Experimental)
  Interventions: Drug: AG013736

INTERVENTIONS:
Drug: AG013736 — AG013736, tablets 5 mg BID daily until tumor progression or toxicity

SUMMARY:
This is a Phase 2 study being conducted at multiple centers in the United States. Patients having thyroid cancer that has spread to other parts of the body (i.e., metastatic) are eligible to participate. Patients must have disease that was not controlled by previous treatment with radioactive iodine (131I) or not be good candidates for such treatment. The purpose of the study is to test whether the angiogenesis inhibitor AG-013736 is an effective treatment for metastatic thyroid cancer as shown by the number of patients in the study who experience significant and durable tumor shrinkage.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented thyroid cancer with metastases.
* Failure of radioactive iodine (131I) to control the disease or radioactive iodine (131I) is not an appropriate therapy (e.g. due to lack of iodine uptake by the tumor)

Exclusion Criteria:

* Central lung lesions involving major blood vessels (arteries or veins).(Central lesions that maintain the structural integrity of vessels have the potential to bleed if the tumor lesion undergoes necrosis. MRI or CT angiography should be used in any case where there is any question as to whether blood vessels are involved.)
* Patients with a history of hemoptysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- [Derived] Cohen EE, Tortorici M, Kim S, Ingrosso A, Pithavala YK, Bycott P. A Phase II trial of axitinib in patients with various histologic subtypes of advanced thyroid cancer: long-term outcomes and pharmacokinetic/pharmacodynamic analyses. Cancer Chemother Pharmacol. 2014 Dec;74(6):1261-70. doi: 10.1007/s00280-014-2604-8. Epub 2014 Oct 15. PMID 25315258
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061014&StudyName=Study%20of%20the%20Anti-angiogenesis%20Agent%20AG-013736%20in%20Patients%20with%20Metastatic%20Thyroid%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: Axitinib (AG-013736) tablet administered orally at a dose of 5 milligram (mg) twice daily (BID) in cycles of 4 weeks. Treatment was administered continuously until progression or unacceptable toxicity occurred or the participant withdrew consent.
Period: Overall Study
Arm/Group | Axitinib
Started | 60
Completed | 0
Not Completed | 60
Not completed — Adverse Event | 11
Not completed — Death | 4
Not completed — Lack of Efficacy | 17
Not completed — Lost to Follow-up | 2
Not completed — progressive disease | 2
Not completed — clinical progression | 1
Not completed — roll-over to another study | 14
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Groups:
- Axitinib: Axitinib (AG-013736) tablet administered orally at a dose of 5 mg BID in cycles of 4 weeks. Treatment was administered continuously until progression or unacceptable toxicity occurred or the participant withdrew consent.
Arm/Group | Axitinib
Number analyzed (Participants) | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed response are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 8 weeks up to 206 weeks
Population: Intent to treat (ITT) population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 60
Percentage of participants | 38.3 [26.1 to 51.8]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time in days from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1). Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline to disease progression or death due to any cause, assessed every 8 weeks up to 206 weeks
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 60
Days | 459 [302 to 610]

3. Secondary Outcome: Duration of Response (DR)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Baseline to disease progression or discontinuation from study due to any cause, assessed every 8 weeks up to 206 weeks
Population: Subgroup of participants from the ITT population with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 23
Days | 625 [382 to 1391]

4. Secondary Outcome: Overall Survival (OS)
Description: Time in days from the start of study treatment to date of death due to any cause. OS was calculated as the death date minus the date of first dose of study medication plus 1. Death was determined from AE data (where outcome was death) or from follow-up contact data (where the participant current status was death). For participants who were alive, overall survival was censored at the last contact.
Time Frame: Baseline to death due to any cause or at least 1 year after the initial dose for the last treated participant
Population: ITT population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 60
Days | 1068 [568 to NA] — Upper limit of confidence interval was not estimable due to the high number of participants censored for survival.

5. Other Pre Specified Outcome: Population Pharmacokinetics for Axitinib (AG-013736) Plasma Concentrations
Description: Population pharmacokinetic analysis involved mixed effects modeling using nonlinear mixed effects modeling (NONMEM) software. The intent of this analysis was to establish a basic population pharmacokinetic model for axitinib (AG-013736) and to determine inter-individual and residual variability in population (oral) clearance, and volume of distribution of drug. Relationship of demographic variables (gender, age, body weight, height and ethnicity), concomitant medications and measures of altered hepatic and renal function were examined by fitting measured axitinib (AG-013736) concentrations.
Time Frame: Day 1 (pre-dose), Day 29, Day 57 and then every 8 weeks up to 206 weeks
Population: Population pharmacokinetic values were not summarized as descriptive statistics since the data was not available for the single study and data for all the axitinib (AG-013736) Phase 2 studies would be pooled together in a separate report.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Axitinib
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Plasma Concentrations of Soluble Proteins
Description: Plasma concentrations of soluble proteins (vascular endothelial growth factor [VEGF], placental growth factor [PlGF] and soluble vascular endothelial growth factor receptor-2 [sVEGFR2]) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity. It is presented as ratio to baseline, which is obtained by dividing the plasma soluble protein concentration at each time point by its concentration at baseline.
Time Frame: Day 1 (pre-dose) and then every 8 weeks up to 206 weeks
Population: Ratio to baseline values for plasma soluble proteins were not summarized as descriptive statistics since the data was not available for the single study and data for all the axitinib Phase 2 studies would be pooled together in a separate report.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Axitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 32/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=60)
Atrial fibrillation (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Conduction disorder, not otherwise specified (NOS) (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Blindness (Eye disorders) | 1
Abdominal pain NOS (Gastrointestinal disorders) | 1
Diarrhoea NOS (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pancreatitis NOS (Gastrointestinal disorders) | 1
Vomiting NOS (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 3
Disease progression NOS (General disorders) | 3
Fall (General disorders) | 1
Fatigue (General disorders) | 1
Granuloma NOS (General disorders) | 1
Multi-organ failure (General disorders) | 1
Neck oedema (General disorders) | 1
Oedema NOS (General disorders) | 1
Pyrexia (General disorders) | 1
Weakness (General disorders) | 1
Gallbladder disorder NOS (Hepatobiliary disorders) | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1
Actinomycotic pulmonary infection (Infections and infestations) | 1
Arthritis infective NOS (Infections and infestations) | 1
Infection NOS (Infections and infestations) | 1
Ludwig angina (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Pneumonia NOS (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 1
Tracheitis NOS (Infections and infestations) | 1
Fractured pelvis NOS (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Bone sarcoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Encephalopathy NOS (Nervous system disorders) | 1
Headache NOS (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Visual field defect NOS (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Airway obstruction NOS (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma aggravated (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory tract haemorrhage NOS (Respiratory, thoracic and mediastinal disorders) | 2
Sweating increased (Skin and subcutaneous tissue disorders) | 1
Deep venous thrombosis NOS (Vascular disorders) | 1
Hyperaemia (Vascular disorders) | 1
Hypertension NOS (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=60)
Anaemia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 5
Tachycardia (Cardiac disorders) | 4
Ear pain (Ear and labyrinth disorders) | 4
Vision blurred (Eye disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 16
Abdominal pain upper (Gastrointestinal disorders) | 12
Cheilitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 40
Dry mouth (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 24
Dysphagia (Gastrointestinal disorders) | 12
Flatulence (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11
Glossodynia (Gastrointestinal disorders) | 6
Haemorrhoids (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 30
Oral pain (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 18
Swollen tongue (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 10
Chills (General disorders) | 12
Disease progression (General disorders) | 3
Fatigue (General disorders) | 42
Mucosal inflammation (General disorders) | 16
Oedema (General disorders) | 6
Oedema peripheral (General disorders) | 15
Pain (General disorders) | 7
Pyrexia (General disorders) | 11
Seasonal allergy (Immune system disorders) | 4
Bronchitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 5
Laryngitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 6
Rhinitis (Infections and infestations) | 11
Sinusitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood glucose increased (Investigations) | 3
Blood potassium decreased (Investigations) | 6
Blood pressure increased (Investigations) | 3
Weight decreased (Investigations) | 24
Decreased appetite (Metabolism and nutrition disorders) | 28
Dehydration (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 11
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 17
Dysgeusia (Nervous system disorders) | 12
Headache (Nervous system disorders) | 27
Hypoaesthesia (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 9
Sciatica (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 15
Haematuria (Renal and urinary disorders) | 6
Pollakiuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 16
Urinary incontinence (Renal and urinary disorders) | 3
Erectile dysfunction (Reproductive system and breast disorders) | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 23
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 11
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 13
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 18
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 3
Hot flush (Vascular disorders) | 3
Hypertension (Vascular disorders) | 28
Hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Population pharmacokinetics and plasma concentrations of soluble proteins were not presented, as the data was not available for the single study and data for all the axitinib (AG-013736) Phase 2 studies would be pooled together in a separate report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.